CLINICAL TRIAL: NCT00005251
Title: Genetic Analysis of Familial Hypertrophic Cardiomyopathy
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1133; R01HL042467 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2000-06

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Myocardial Diseases; Cardiomyopathy, Hypertrophic
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Cardiomyopathies; Cardiomyopathy, Hypertrophic

SUMMARY:
To map the genetic defect responsible for familial hypertrophic cardiomyopathy.

DETAILED DESCRIPTION:
BACKGROUND:

Familial hypertrophic cardiomyopathy is a disease of heart muscle that is genetically transmitted as an autosomal dominant trait, with a high degree of penetrance. Affected individuals typically have asymmetric thickening of the interventricular septum often involving the adjacent left ventricular free wall. Histologically, myocardial cells are enlarged and muscle bundles are grossly disorganized, producing a whorled pattern. The physiologic consequence of this cardiomyopathy is diastolic dysfunction with impaired ventricular relaxation and elevated diastolic pressures in the heart and pulmonary vasculature. Patients can experience dyspnea, angina, palpitations, and syncope. Complications of the disease include atrial fibrillation, congestive heart failure, thromboembolism, and most importantly, sudden death.

DESIGN NARRATIVE:

The three kindreds studied included one in Iceland, one in the St. Lawrence region in Canada, and one in the Pittsburgh, Pennsylvania area. Pedigrees were established for the three kindreds. All family members were clinically evaluated by physical exam, electrocardiogram, and comprehensive M-mode and two-dimensional echocardiography. Lymphoblastoid cell lines were derived from all members of the three pedigrees. Restriction fragment length polymorphism analyses were used to identify a DNA probe that was linked to familial hypertrophic cardiomyopathy. Studies were conducted to determine if the familial hypertrophic cardiomyopathy locus was the same in all three kindreds and to identify the gene responsible.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1990-01; Study Completion 1995-03 (Actual)

REFERENCES:
- [Background] Watkins H, Thierfelder L, Hwang DS, McKenna W, Seidman JG, Seidman CE. Sporadic hypertrophic cardiomyopathy due to de novo myosin mutations. J Clin Invest. 1992 Nov;90(5):1666-71. doi: 10.1172/JCI116038. PMID 1430197
- [Background] Watkins H, Seidman CE, MacRae C, Seidman JG, McKenna W. Progress in familial hypertrophic cardiomyopathy: molecular genetic analyses in the original family studied by Teare. Br Heart J. 1992 Jan;67(1):34-8. doi: 10.1136/hrt.67.1.34. No abstract available. PMID 1739523
- [Background] Seidman CE, Seidman JG. Mutations in cardiac myosin heavy chain genes cause familial hypertrophic cardiomyopathy. Mol Biol Med. 1991 Apr;8(2):159-66. PMID 1806760
- [Background] Solomon SD, Jarcho JA, McKenna W, Geisterfer-Lowrance A, Germain R, Salerni R, Seidman JG, Seidman CE. Familial hypertrophic cardiomyopathy is a genetically heterogeneous disease. J Clin Invest. 1990 Sep;86(3):993-9. doi: 10.1172/JCI114802. PMID 1975599
- [Background] Geisterfer-Lowrance AA, Kass S, Tanigawa G, Vosberg HP, McKenna W, Seidman CE, Seidman JG. A molecular basis for familial hypertrophic cardiomyopathy: a beta cardiac myosin heavy chain gene missense mutation. Cell. 1990 Sep 7;62(5):999-1006. doi: 10.1016/0092-8674(90)90274-i. PMID 1975517
- [Background] Solomon SD, Geisterfer-Lowrance AA, Vosberg HP, Hiller G, Jarcho JA, Morton CC, McBride WO, Mitchell AL, Bale AE, McKenna WJ, et al. A locus for familial hypertrophic cardiomyopathy is closely linked to the cardiac myosin heavy chain genes, CRI-L436, and CRI-L329 on chromosome 14 at q11-q12. Am J Hum Genet. 1990 Sep;47(3):389-94. PMID 1975475
- [Background] Tanigawa G, Jarcho JA, Kass S, Solomon SD, Vosberg HP, Seidman JG, Seidman CE. A molecular basis for familial hypertrophic cardiomyopathy: an alpha/beta cardiac myosin heavy chain hybrid gene. Cell. 1990 Sep 7;62(5):991-8. doi: 10.1016/0092-8674(90)90273-h. PMID 2144212
- [Background] Knowlton KU, Rockman HA, Itani M, Vovan A, Seidman CE, Chien KR. Divergent pathways mediate the induction of ANF transgenes in neonatal and hypertrophic ventricular myocardium. J Clin Invest. 1995 Sep;96(3):1311-8. doi: 10.1172/JCI118166. PMID 7657806
- [Background] Watkins H, MacRae C, Thierfelder L, Chou YH, Frenneaux M, McKenna W, Seidman JG, Seidman CE. A disease locus for familial hypertrophic cardiomyopathy maps to chromosome 1q3. Nat Genet. 1993 Apr;3(4):333-7. doi: 10.1038/ng0493-333. PMID 7981753
- [Background] Thierfelder L, Watkins H, MacRae C, Lamas R, McKenna W, Vosberg HP, Seidman JG, Seidman CE. Alpha-tropomyosin and cardiac troponin T mutations cause familial hypertrophic cardiomyopathy: a disease of the sarcomere. Cell. 1994 Jun 3;77(5):701-12. doi: 10.1016/0092-8674(94)90054-x. PMID 8205619
- [Background] Anan R, Greve G, Thierfelder L, Watkins H, McKenna WJ, Solomon S, Vecchio C, Shono H, Nakao S, Tanaka H, et al. Prognostic implications of novel beta cardiac myosin heavy chain gene mutations that cause familial hypertrophic cardiomyopathy. J Clin Invest. 1994 Jan;93(1):280-5. doi: 10.1172/JCI116957. PMID 8282798
- [Background] Watkins H, Thierfelder L, Anan R, Jarcho J, Matsumori A, McKenna W, Seidman JG, Seidman CE. Independent origin of identical beta cardiac myosin heavy-chain mutations in hypertrophic cardiomyopathy. Am J Hum Genet. 1993 Dec;53(6):1180-5. PMID 8250038
- [Background] Solomon SD, Wolff S, Watkins H, Ridker PM, Come P, McKenna WJ, Seidman CE, Lee RT. Left ventricular hypertrophy and morphology in familial hypertrophic cardiomyopathy associated with mutations of the beta-myosin heavy chain gene. J Am Coll Cardiol. 1993 Aug;22(2):498-505. doi: 10.1016/0735-1097(93)90055-6. PMID 8335820
- [Background] Watkins H, Rosenzweig A, Hwang DS, Levi T, McKenna W, Seidman CE, Seidman JG. Characteristics and prognostic implications of myosin missense mutations in familial hypertrophic cardiomyopathy. N Engl J Med. 1992 Apr 23;326(17):1108-14. doi: 10.1056/NEJM199204233261703. PMID 1552912